CLINICAL TRIAL: NCT00652665
Title: To Compare the Relative Bioavailability of Leflunomide 20mg Tablets (Kali) With That of ARAVA 20mg Tablets(Aventis) Under Fasting Conditions
Brief Title: Bioavailability Study of Leflunomide Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Dr. Alfred Elvin/ Director Biopharmaceutics, Par Pharmaceutical, Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B033201
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-03

CONDITIONS: To Determine the Bioequivalence Study Under Fasting
Keywords: Bioequivalence, single-dose, fasting
MeSH Terms: conditions — Fasting | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Subjects received kali product under fasting conditions
  Interventions: Drug: Leflunomide
- B (Active Comparator): Subjects received Aventis product under fasting conditions
  Interventions: Drug: ARAVA

INTERVENTIONS:
Drug: Leflunomide — Tablets, 20mg, single-dose
  Other Names: ARAVA
  Arms: A
Drug: ARAVA — Tablets, 20mg,single-dose
  Other Names: Leflunomide
  Arms: B

SUMMARY:
To compare the single-dose Bioavailability of Kali and Aventis

DETAILED DESCRIPTION:
To compare the relative Bioavailability of leflunomide 20mg tablets with that of ARAVA 20mg tablets in healthy, adult subjects under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be at least 18 years of age.
* Females must be physically unable to become pregnant.
* Males must be vasectomized.
* Each subject shall be given a general physical examination within 28 days of initiation of the study.
* Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre- study screening process
* At the end of study, the subject will have an exit evaluation consisting of interim history, global evaluation, clinical laboratory measurements
* Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements
* Clinical laboratory measurements will include hematology, clinical chemistry, urine analysis, HIV screen, hepatitis-B,C screen, drugs of abuse screen before dosing.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction,or recent serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study
* Subjects whose clinical laboratory test values are greater tahn 20% outside the normal range may be retested.If the clinical values are out side the range on retesting the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.Subjects who have a history of allergic responses to cholestyramine should be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs and abuse as part of the clinical laboratory screening procedures and at check-in before dosing. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty(30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty(30)days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant or who are able(women with child bearing potential) to become pregnant during the study will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in. Subjects with positive or inconclusive results will be withdrawn from the study.
* Male subjects who are physically able to father a child will not be allowed to participate. Male subjects must be vasectomized(at least 3 months) with medical verification.
* Subjects who have taken any product containing leflunomide within 180 days of dosing will not be allowed to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Hong, Principal Investigator — Novum Pharmaceutical Research Services